CLINICAL TRIAL: NCT05789576
Title: A Phase 4, Open-label Study to Investigate the Efficacy and Safety of VTAMA® (Tapinarof) Cream, 1% in the Treatment of Plaque Psoriasis Occurring in the Head and Neck Region
Brief Title: A Study to Investigate Efficacy and Safety of VTAMA® (Tapinarof) Cream, 1% in Plaque Psoriasis in the Head and Neck Region
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-4002
Record Dates: First submitted 2023-03-14; First posted 2023-03-29 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-08

CONDITIONS: Psoriasis
Keywords: Tapinarof; Plaque Psoriasis; Scalp Psoriasis; Psoriasis; Phase 4; Topical; Open-label; Efficacy; Safety; Adult; Face Psoriasis; Neck Psoriasis; Psoriatic conditions
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VTAMA (tapinarof) cream, 1% (Experimental): VTAMA (tapinarof) cream, 1% applied topically once daily
  Interventions: Drug: VTAMA (tapinarof) cream, 1%

INTERVENTIONS:
Drug: VTAMA (tapinarof) cream, 1% — VTAMA (tapinarof) cream, 1% applied topically once daily
  Other Names: DMVT-505

SUMMARY:
This is an open-label, multi-center study to evaluate the efficacy and safety of VTAMA (tapinarof) cream, 1% in adults with plaque psoriasis occurring in the head and neck region

DETAILED DESCRIPTION:
This is an open-label study in which participants with plaque psoriasis in the head and neck region will be assigned to receive VTAMA (tapinarof) cream, 1% once daily for 12 weeks. Study participants will have a follow-up period of 1 week. The study duration will be up to 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, at the time of signing the informed consent
* Participants with clinical diagnosis of plaque psoriasis, including lesion(s) in the head and neck region and stable disease in the head and neck region for at least 3 months prior to the study
* Participant has a plaque psoriasis lesion in the head and neck region that is suitable for evaluation as the target lesion and has a PGA (target lesion) score of 2 (Mild), 3 (Moderate), or 4 (Severe) at Screening and Baseline
* Female subjects of child bearing potential who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study
* Negative pregnancy test at Baseline (Day 1)
* Capable of giving written informed consent

Exclusion Criteria:

* Diagnosis of a type of psoriasis other than plaque psoriasis
* Any sign of infection of any of the psoriatic lesions
* Concurrent significant dermatologic or inflammatory condition other than plaque psoriasis that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
* History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with participation in the study and ability to understand and give informed consent
* History of sensitivity to the study product, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation in the study
* Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001); previous or current use of VTAMA® (Tapinarof) cream, 1%
* Use of any prohibited medication or procedure within the indicated period before the baseline visit including other investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer)
* UV light therapy or prolonged exposure to natural or artificial sources of UV radiation (e.g., phototherapy, tanning beds/booths, or therapeutic sunbathing) within 4 weeks prior to the Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Dermavant Investigative Site, Macon, Georgia
  - Dermavant Investigative Site, Chicago, Illinois
  - Dermavant Investigative Sites, Rockville, Maryland
  - Dermavant Investigative Site, Auburn Hills, Michigan
  - Dermavant Investigative Site, Detroit, Michigan
  - Dermavant Investigative Site, Las Vegas, Nevada
  - Dermavant Investigative Site, Portsmouth, New Hampshire
  - Dermavant Investigative Site, Kew Gardens, New York
  - Dermavant Investigative Site, Marion, Ohio
  - Dermavant Investigative Site, Arlington, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VTAMA (Tapinarof) Cream, 1%
Started | 31
Completed | 24
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | VTAMA (Tapinarof) Cream, 1%
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (16.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 31
PGA (Target Lesion) [Count of Participants; unit: Participants]
  0 - Clear | 0
  1 - Almost Clear | 0
  2 - Mild | 12
  3 - Moderate | 17
  4 - Severe | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a Target Lesion Physician Global Assessment (PGA) Score in the Head and Neck Region of Clear (0) or Almost Clear (1) With a ≥ 2-grade Improvement
Description: Physician Global Assessment (PGA) is a clinical tool for assessing the current state/severity of a participant's psoriasis in a target lesion of the head and neck region at a given timepoint. It is a static 5-point assessment of plaque qualities on the clinical characteristics of erythema, scaling, and plaque thickness/elevation within the head and neck region. The PGA ranges from 0 to 4, and is assessed as Clear (0), Almost Clear (1), Mild (2), Moderate (3), and Severe (4). Higher PGA scores represent more severe disease.
Time Frame: from Baseline to Week 12
Population: Observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | VTAMA (Tapinarof) Cream, 1%
Number analyzed (Participants) | 26
Participants | 23

2. Secondary Outcome: Time to Achieve a Target Lesion PGA Score of Clear (0) or Almost Clear (1) With a ≥ 2-grade Improvement
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Observed cases
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | VTAMA (Tapinarof) Cream, 1%
Number analyzed (Participants) | 31
days | 29.0 [15.00 to 53.00]

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | VTAMA (Tapinarof) Cream, 1%
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 18/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTAMA (Tapinarof) Cream, 1% (N=31)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTAMA (Tapinarof) Cream, 1% (N=31)
Folliculitis (Infections and infestations) | 6 (6)
Sinusitis (Infections and infestations) | 2 (2)
Seborrheic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05789576/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT05789576/SAP_001.pdf